CLINICAL TRIAL: NCT03782077
Title: Effect of Deflation of Pneumatic Tourniquet on the Change of Optic Nerve Sheath Diameter in Patients Undergoing Knee Surgery
Brief Title: Change of Optic Nerve Sheath Diameter After Deflation of Pneumatic Tourniquet
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hajung Kim, Clinical instructor, Asan Medical Center
Other Study IDs: 2018-1172
Record Dates: First submitted 2018-12-19; First posted 2018-12-20 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Intracranial Pressure Increase
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Deflation of pneumatic tourniquet — Deflation of pneumatic tourniquet

SUMMARY:
The purpose of this study is to evaluate the change of the optic nerve sheath diameter after deflation of pneumatic tourniquet.

DETAILED DESCRIPTION:
Deflation of pneumatic tourniquet could induces many changes in various organ systems. It has been shown to affect intracranial pressure. Thus, the investigators evaluate the change of optic nerve sheath diameter using ultrasound after deflation of pneumatic tourniquet in patients undergoing knee surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1-4
* patients undergoing knee surgery using pneumatic tourniquet

Exclusion Criteria:

* patients who refuse to participate in this study
* patients with history of cerebrovascular disease
* patients who are judged ineligible by the medical staff to participate in the study for other reasons

Ages: 18 Years to 79 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing knee surgery using pneumatic tourniquet
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2018-12-13 (Actual)

PRIMARY OUTCOMES:
change of optic nerve sheath diameter | 5 minutes before deflation and at 5-minute intervals for 10 minutes after deflation
  difference in optic nerve sheath diameter measured using ultrasound before and after deflation of pneumatic tourniquet

CONTACTS AND LOCATIONS:
Overall Officials: Won Uk Koh, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim HJ, Kim YJ, Kim J, Kim H, Ro YJ, Koh WU. Change in the optic nerve sheath diameter after deflation of a pneumatic tourniquet: a prospective observational study. Sci Rep. 2022 Jan 11;12(1):521. doi: 10.1038/s41598-021-04457-4. PMID 35017581